CLINICAL TRIAL: NCT03289910
Title: NCI 10147: A Phase II Randomized Study of Topotecan/Carboplatin With or Without Veliparib in Advanced Myeloproliferative Disorders and Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Topotecan Hydrochloride and Carboplatin With or Without Veliparib in Treating Advanced Myeloproliferative Disorders and Acute Myeloid Leukemia or Chronic Myelomonocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2017-01715; NCI-2017-01715 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ETCTN10147; 10147 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10147 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-21 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Atypical Chronic Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Essential Thrombocythemia; Myelodysplastic/Myeloproliferative Neoplasm; Myelofibrosis; Polycythemia Vera; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Myelodysplastic-Myeloproliferative Diseases; Primary Myelofibrosis; Polycythemia Vera | interventions — Carboplatin; Topotecan; veliparib

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (veliparib, topotecan hydrochloride, carboplatin) (Experimental): Patients receive veliparib PO BID on days 1-21 and topotecan hydrochloride IV continuously over 24 hours and carboplatin IV continuously over 24 hours on days 3-7. Treatment repeats every 28-63 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Topotecan; Drug: Topotecan Hydrochloride; Drug: Veliparib
- Arm B (topotecan hydrochloride, carboplatin) (Active Comparator): Patients receive topotecan hydrochloride IV continuously over 24 hours and carboplatin IV continuously over 24 hours on days 1-5. Treatment repeats every 28-63 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Topotecan; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888
  Arms: Arm A (veliparib, topotecan hydrochloride, carboplatin)

SUMMARY:
This phase II trial studies how well topotecan hydrochloride and carboplatin with or without veliparib work in treating patients with myeloproliferative disorders that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced), and acute myeloid leukemia or chronic myelomonocytic leukemia. Drugs used in chemotherapy, such as topotecan hydrochloride and carboplatin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Veliparib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving topotecan hydrochloride, carboplatin, and veliparib may work better in treating patients with myeloproliferative disorders and acute myeloid leukemia or chronic myelomonocytic leukemia compared to topotecan hydrochloride and carboplatin alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate and compare the complete response/complete response with incomplete recovery (CR/CRi) rate of induction therapy with topotecan hydrochloride (topotecan)/carboplatin (T/C) with or without veliparib (V) in myeloproliferative disorder associated leukemias and chronic myelomonocytic leukemia (CMML).

SECONDARY OBJECTIVES:

I. To evaluate and compare the toxicities of T/C/V versus (vs.) T/C. II. To compare the 2-year disease-free survival (DFS) and overall survival (OS) in response to T/C/V vs. T/C.

III. To detect and compare the presence of minimal residual disease (MRD) remaining after T/C/V vs. T/C.

IV. Evaluate predictive biomarkers of response via assessment of pretreatment impaired homologous recombination via assessment of:

IVa. Next generation sequencing (NGS) panel for genes mutated in myeloid malignancies done as standard of care per institution.

IVb. Functional impairment of deoxyribonucleic acid (DNA) damage response via assessment of pretreatment samples for radiation-induced RAD51 foci.

IVc. Topotecan-induced stabilization of topoisomerase I-DNA covalent complexes, which has recently been observed to be a critical predictor of response to combination of a topoisomerase I poison and PARP inhibitor in xenografts.

V. To evaluate veliparib exposure and contribution to response (efficacy and toxicity).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive veliparib orally (PO) twice daily (BID) on days 1-21 and topotecan hydrochloride intravenously (IV) continuously over 24 hours and carboplatin IV continuously over 24 hours on days 3-7. Treatment repeats every 28-63 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive topotecan hydrochloride IV continuously over 24 hours and carboplatin IV continuously over 24 hours on days 1-5. Treatment repeats every 28-63 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for a minimum of 30 days, or longer.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA
* Newly diagnosed acute myeloid leukemia (AML) associated with antecedent myeloproliferative disorder (polycythemia vera, essential thrombocythemia, myelofibrosis, atypical chronic myeloid leukemia, chronic myelomonocytic leukemia and related undifferentiated myeloproliferative/myelodysplastic disorders)
* Relapsed/refractory AML associated with antecedent myeloproliferative disorder (polycythemia vera, essential thrombocythemia, myelofibrosis, atypical chronic myeloid leukemia, chronic myelomonocytic leukemia and related undifferentiated myeloproliferative/myelodysplastic disorders) who have received two or fewer prior induction chemotherapy courses
* Accelerated phase myeloproliferative disorders per Zeider et al with two or fewer prior therapies

  * For aggressive phase myeloproliferative disorders (MPD) (polycythemia vera, essential thrombocythemia, Philadelphia [Ph]-negative chronic myelogenous leukemia), one or more of the following criteria must be met: marrow blasts > 5%, peripheral blood blasts plus progranulocytes > 10%, new onset or increasing myelofibrosis, new onset or > 25% increase in hepatomegaly or splenomegaly, new onset constitutional symptoms (fever, weight loss, splenic pain, bone pain). Zeider et al
  * For chronic myelomonocytic leukemia (CMML), the following criteria must be met: 5-19% bone marrow blasts (aggressive) or >= 20% marrow blasts (transformation)
* Bone marrow and/or peripheral blood specimens will be submitted for correlative studies; patients with a dry tap will still be eligible
* RANDOMIZATION ELIGIBILITY CRITERIA
* Bone marrow aspirate and/or peripheral blood specimens were submitted to the central lab and site has confirmation by the local institution that the patient meets one of the criteria specified above
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 or Karnofsky >= 60%
* Total bilirubin less than 2.0 mg/dL unless due to Gilbert's syndrome, then less than 5.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) less than 5 x institutional upper limit of normal
* Creatinine clearance glomerular filtration rate (GFR) greater than 30 ml/min per modified Cockcroft-Gault formula
* Interval of greater than 4 weeks since allogeneic blood or marrow transplantation (BMT) if performed; and absence of active graft versus host disease (GVHD)
* The effects of veliparib on the developing human fetus are unknown; for this reason and because PARP inhibiting agents as well as topoisomerase inhibitors and platinating agents are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months following the last dose of study drug; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of veliparib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study with the exception of hydroxyurea for cytoreduction; therapy with tyrosine kinase inhibitors (TKIs) directed against JAK2, BCR-ABL or FLT3 will be allowed to be continued until 24 hours prior to start of therapy on trial
* Patients with active uncontrolled infection; antibiotic therapy for fevers, and continuation of treatment of prior infection are allowed
* Patients who have active central nervous system (CNS) disease are excluded; patients with known active CNS leukemia should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients who are receiving any other investigational agents; patients who have completed therapy with an investigational agent should be off this therapy for at least 5 half-lives or two weeks, whichever is shorter
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib, topotecan or carboplatin
* Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because veliparib is PARP inhibiting agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with veliparib, breastfeeding should be discontinued if the mother is treated with veliparib; these potential risks may also apply to topotecan and carboplatin used in this study
* Human immunodeficiency virus (HIV)-patients positive patients are not excluded if they have CD4+ cells >= 250/mm^3 and negligible viral load and are on a stable combination antiretroviral therapy
* History of uncontrolled seizure disorder, including focal or generalized seizure within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2025-12-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Keith W Pratz, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (6):
- United States (6):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Richardson DR, Green SD, Foster MC, Zeidner JF. Secondary AML Emerging After Therapy with Hypomethylating Agents: Outcomes, Prognostic Factors, and Treatment Options. Curr Hematol Malig Rep. 2021 Feb;16(1):97-111. doi: 10.1007/s11899-021-00608-6. Epub 2021 Feb 20. PMID 33609248

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Started | 16 | 9
Completed | 16 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin) | Total
Number analyzed (Participants) | 16 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 8 | 5 | 13
Age, Continuous [Median (Full Range); unit: years] | 65 [33 to 75] | 69 [46 to 74] | 66 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 8 | 24
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Based on published standards for acute leukemias, Complete Response (CR) means less than 5% leukemic blasts in the bone marrow, no blasts in the blood, no longer presence of cytogenetic abnormalities, no longer presence of extramedullary disease, with or without absolute neutrophil count or platelet count recovery; Partial Remission (PR) includes the criteria for Complete Remission except there are 5-25% leukemic blasts in the bone marrow and there is absolute neutrophil count and platelet count recovery; Hematologic Improvement (HI) means the disease has not gotten worse and there is at least a 20% decrease in the leukemic blasts in the bone marrow and/or a decrease in leukemia symptoms. Response = CR, PR, or HI.
Time Frame: Up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 16 | 9
Participants
  Participants with a response | 5 | 4
  Participants who did not have a response | 11 | 5

2. Secondary Outcome: The Highest Grade Adverse Event Experienced
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 16 | 9
Participants
  Grade 5 Adverse Events | 0 | 1
  Grade 4 Adverse Events | 14 | 8
  Grade 3 Adverse Events | 2 | 0

3. Secondary Outcome: Number of Participants Without Disease at Study Completion
Description: Study completion was either death or completion of all protocol-specified activities, whichever came first. Participants who came off study due to disease-related death were counted as having disease.
Time Frame: Up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 16 | 9
Participants | 3 | 3

4. Secondary Outcome: Duration of Disease-free Survival
Description: Disease-free survival is defined as participants who are still alive and without disease at study completion. Study completion was either death or completion of all protocol-specified activities, whichever came first.
Time Frame: Up to 7 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 16 | 9
days | 120 [37 to 137] | 89 [27 to 137]

5. Secondary Outcome: Number of Participants Still Alive at Study Completion
Description: Study completion was either death or completion of all protocol-specified activities, whichever came first.
Time Frame: Up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 16 | 9
Participants | 5 | 5

6. Secondary Outcome: Duration of Overall Survival at the Time of Study Completion
Description: Study completion was either death or completion of all protocol-specified activities, whichever came first. Duration was measured from the date of registration to the participant's study completion date.
Time Frame: Up to 7 months
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 16 | 9
Days | 83 [74 to 295] | 123 [82 to 295]

7. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD) After Treatment
Description: Minimal residual disease (MRD) refers to a small number of leukemic cells that remain after treatment.
Time Frame: Up to 7 months
Population: Data was not collected.
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Distribution of Mutations in Deoxyribonucleic Acid (DNA) Repair Defects Via Assessment in Leukemia Mutation Panel
Description: Will be summarized using descriptive statistics. The association response will be described with appropriate tests for continuously measured biomarkers (t tests, Wilcoxon rank sum tests) and categorical biomarkers (Fisher's exact test). Descriptive analyses will be performed for the whole cohort and also separately for Arms A and B. Differential treatment outcomes for patient subgroups may be explored using appropriate tests for interactions.
Time Frame: Baseline
Population: Data not collected.
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Frequency of Patients With Functional Impairment of DNA Damage Response Via Assessment With RAD51 Assay
Description: Will be reported with exact binomial 95% confidence intervals. The association response will be described with appropriate tests for continuously measured biomarkers (t tests, Wilcoxon rank sum tests) and categorical biomarkers (Fisher's exact test). Descriptive analyses will be performed for the whole cohort and also separately for Arms A and B. Differential treatment outcomes for patient subgroups may be explored using appropriate tests for interactions.
Time Frame: Baseline
Population: Data not collected.
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Topotecan-induced Stabilization of Topoisomerase I-DNA Covalent Complexes
Description: Topotecan-induced stabilization of topoisomerase I-DNA covalent complexes from peripheral blood
Time Frame: Up to 7 months
Population: Data not collected.
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Pharmacokinetic Sampling Studies Measured Using a Validated Liquid Chromatography/Tandem Mass Spectrometric Method in Plasma and Bone Marrow
Description: Plasma trough levels will be obtained weekly through the first cycle to provide a steady-state assessment. Steady-state plasma concentrations will be calculated for each patient. Exploratory correlative studies between veliparib exposure (plasma and bone marrow) with pharmacodynamic (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics. Significance for comparisons will be at the p < 0.05 level.
Time Frame: Pre-treatment, day 1, day 8, day 14, day 15, and day 22 (approximately 24 hours post last dose)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up 7 months
Arm/Group | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) | Arm B (Topotecan Hydrochloride, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 11/16 | 4/9
Serious Adverse Events (participants affected / at risk) | 4/16 | 4/9
Other Adverse Events (participants affected / at risk) | 16/16 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) (N=16) | Arm B (Topotecan Hydrochloride, Carboplatin) (N=9)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Cardiac troponin I increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Veliparib, Topotecan Hydrochloride, Carboplatin) (N=16) | Arm B (Topotecan Hydrochloride, Carboplatin) (N=9)
Anemia (Blood and lymphatic system disorders) | 14 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 5
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 6 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
mild bleeding (Ear and labyrinth disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 1
mild L subconjunctival hemorrhage (Eye disorders) | 0 | 1
Right eye drainage (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 11 | 4
Anal mucositis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 3 | 0
Belching (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 4
Colitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 13 | 9
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
enteritis (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
GI bleed, site unknown (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 10 | 7
Oral hemorrhage (Gastrointestinal disorders) | 2 | 0
Oral pain (Gastrointestinal disorders) | 3 | 1
pneumatosis (Gastrointestinal disorders) | 0 | 1
Rectal fissure (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal pain (Gastrointestinal disorders) | 1 | 0
Small intestinal mucositis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 9 | 5
Chills (General disorders) | 4 | 1
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 5 | 3
Edema trunk (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 8 | 7
Fever (General disorders) | 7 | 3
Generalized edema (General disorders) | 3 | 1
Hypothermia (General disorders) | 0 | 1
Localized edema (General disorders) | 1 | 1
Pain (General disorders) | 5 | 3
cholelithiasis (Hepatobiliary disorders) | 1 | 0
liver parenchyma disease (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 1 | 0
C Reactive Protein > ULN (Immune system disorders) | 0 | 1
Erythrocyte Sedimentation Rate > ULN (Immune system disorders) | 0 | 1
Spleen Disorder (Immune system disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Bilateral nodules (Infections and infestations) | 1 | 0
Bilateral pulmonary nodules (Infections and infestations) | 0 | 1
Bone infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 1
Endocarditis infective (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 4 | 2
Mucosal infection (Infections and infestations) | 0 | 1
multi organ bacteremia (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Salivary gland infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 0
Skin infection (Infections and infestations) | 2 | 2
Soft tissue infection (Infections and infestations) | 1 | 0
Strep salivarious infection (Infections and infestations) | 1 | 0
Thrush (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 2
Alanine aminotransferase increased (Investigations) | 8 | 5
Alkaline phosphatase increased (Investigations) | 11 | 4
Aspartate aminotransferase increased (Investigations) | 10 | 3
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 12 | 3
Blood lactate dehydrogenase increased (Investigations) | 1 | 3
Creatinine increased (Investigations) | 6 | 1
D Dimer Increased (Investigations) | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 2
Fibrinogen decreased (Investigations) | 2 | 0
GGT increased (Investigations) | 1 | 0
Haptoglobin decreased (Investigations) | 0 | 1
INR increased (Investigations) | 2 | 3
Left inguinal hernia (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Liver Abscess (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 16 | 8
Neutrophil count decreased (Investigations) | 14 | 7
Platelet count decreased (Investigations) | 15 | 8
Swollen scrotum (Investigations) | 0 | 1
Weight loss (Investigations) | 3 | 6
White blood cell count increased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 16 | 9
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 9 | 6
early satiety (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hypernatremia (Metabolism and nutrition disorders) | 5 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 8 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 15 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 3
Hyponatremia (Metabolism and nutrition disorders) | 10 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 10 | 5
post-prandial discomfort (Metabolism and nutrition disorders) | 1 | 0
vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3
R toenail changes (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 4
Dysgeusia (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 4 | 2
Hypersomnia (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 3 | 1
Tremor (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Confusion (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Glucosuria (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 6 | 1
Proteinuria (Renal and urinary disorders) | 4 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2
tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hives (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 3
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 9 | 4
Hypotension (Vascular disorders) | 6 | 3
Thromboembolic event (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT03289910/Prot_SAP_000.pdf